CLINICAL TRIAL: NCT01783158
Title: Chromoendoscopy to Detect Early Synchronous Second Primary Esophageal Carcinoma in Patients With Squamous Cell Carcinomas of the Head and Neck?
Brief Title: Chromoendoscopy to Detect Early Synchronous Second Primary Esophageal Carcinoma
Acronym: HNSCC
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: RVO-FNOs/2012
Record Dates: First submitted 2013-01-23; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Squamous Cell Carcinomas of the Head and Neck
Keywords: head and neck carcinoma; chromoendoscopy; Lugol's solution; esophageal carcinoma; synchronous tumors; deglutition; deglutition disorders; Newly diagnosed HNSCC
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders | interventions — Esophagoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic group: A total of 132 patients with HNSCC were enrolled in this study. The patients underwent esophagoscopy and chromoendoscopy. The most frequent primary tumors were oropharyngeal (49/132), tumors of the oral cavity (36/132) and larynx (35/132). The majority of subjects (107/132 patients, 81.1%) had advanced HNSCC carcinomas (stages III and IV). Multiple LVLs were discovered in 24 subjects (18.2%), and no LVLs in 108 (81.8%) subjects. Fifty-five LVL biopsy specimens were obtained and assessed. Squamous cell carcinomas were detected in two patients, peptic esophagitis in 11 patients, gastric heterotopic mucosa in two patients, hyperplasia in two patients, and low- and high-grade dysplasia in three patients.
  Interventions: Procedure: Esophagoscopy and chromoendoscopy

INTERVENTIONS:
Procedure: Esophagoscopy and chromoendoscopy — Esophagoscopy - examination of the interior of the esophagus by means of an esophagoscope.
  Chromoendoscopy - a method, which involves the topical application of stains or pigments to improve tissue localization, characterization, or diagnosis during endoscopy.

SUMMARY:
Patients with HNSCC represent a high-risk group for the development of SESCC. Thus, esophagogastrofibroscopy should be performed to detect possible synchronous esophageal carcinomas in these patients.

Although only two patients with synchronous primary carcinomas were found among the patients with newly diagnosed HNSCC in this study, esophagoscopy and better some of advanced endoscopic methods should be recommended after detection of HNSCC to exclude secondary esophageal carcinoma or dysplasia. Staining of the esophagus with Lugol's solution is an easy and inexpensive option and can be done in most of gastroenterology offices.

DETAILED DESCRIPTION:
ABSTRACT Objective: To evaluate the use of flexible esophagoscopy and chromoendoscopy with Lugol's solution in the detection of early esophageal carcinomas (second primary carcinomas) in patients with squamous cell carcinoma of the head and neck (HNSCC).

Methods: All patients with newly diagnosed HNSCC underwent office-based Lugol chromoendoscopy. After flexible esophagoscopy with white light, 3.0% Lugol iodine solution was sprayed over the entire esophageal mucosa. Areas with less-intense staining (LVLs) were evaluated and biopsies taken.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with head and neck carcinoma
* Age 18-65

Exclusion Criteria:

* Recurrent head and neck carcinomas
* Previously diagnosed oesophageal cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed head and neck carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2004-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To detect early synchronous second primary esophageal carcinoma | The primary measure was assessed immediately after the completion of the study by individual patients.
  To evaluate the use of flexible esophagoscopy and chromoendoscopy with Lugol's solution in the detection of early esophageal carcinomas (second primary carcinomas) in patients with squamous cell carcinoma of the head and neck (HNSCC).
  All patients with newly diagnosed HNSCC underwent office-based Lugol chromoendoscopy. After flexible esophagoscopy with white light, 3.0% Lugol iodine solution was sprayed over the entire esophageal mucosa. Areas with less-intense staining (LVLs) were evaluated and biopsies taken.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kominek, MD, PhD, MSc, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia

REFERENCES:
- [Background] Muto M, Hironaka S, Nakane M, Boku N, Ohtsu A, Yoshida S. Association of multiple Lugol-voiding lesions with synchronous and metachronous esophageal squamous cell carcinoma in patients with head and neck cancer. Gastrointest Endosc. 2002 Oct;56(4):517-21. doi: 10.1067/mge.2002.128104. PMID 12297767
- [Background] SLAUGHTER DP, SOUTHWICK HW, SMEJKAL W. Field cancerization in oral stratified squamous epithelium; clinical implications of multicentric origin. Cancer. 1953 Sep;6(5):963-8. doi: 10.1002/1097-0142(195309)6:53.0.co;2-q. No abstract available. PMID 13094644
- [Background] Fukuhara T, Hiyama T, Tanaka S, Oka S, Yoshihara M, Arihiro K, Chayama K. Characteristics of esophageal squamous cell carcinomas and lugol-voiding lesions in patients with head and neck squamous cell carcinoma. J Clin Gastroenterol. 2010 Feb;44(2):e27-33. doi: 10.1097/MCG.0b013e3181b31325. PMID 19730116